CLINICAL TRIAL: NCT02118558
Title: Negative Pressure Wound Therapy -PREVENA in Prevention of Infections After Total Knee Arthroplasty (TKA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0020-14-HMO-CTIL
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Total Knee Replacement
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Negative Pressure Wound Therapy (NPWT) (Experimental)
  Interventions: Device: Negative Pressure Wound Therapy (NPWT)
- standard prophylactic therapy (Active Comparator)
  Interventions: Drug: standard prophylactic therapy

INTERVENTIONS:
Device: Negative Pressure Wound Therapy (NPWT)
  Arms: Negative Pressure Wound Therapy (NPWT)
Drug: standard prophylactic therapy — administration of antibiotics before the first incision, keeping the surgery field sterile and performing several rinsing
  Arms: standard prophylactic therapy

SUMMARY:
This trial is a prospective, single center, unblinded, randomized, controlled study to assess the safety and efficacy of negative pressure wound therapy in preventing infections after TKA surgery . The study will enroll 316 patients that will undergo TKA. patients will be randomized to the treatment group and undergo the study intervention - (NPWT) The intervention will take place at the end of the surgery. The Patients that are randomized to the control group will receive standard treatment. Both groups will be assessed at two weeks and six weeks. period.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18 to 80
* Males- not involved in active military duty.
* Females-non child bearing potential, or females of child-bearing potential who have a negative pregnancy test (hCG urine) within 72 hours of informed consent.

Exclusion Criteria:

* Active systemic or local infection.
* History of malignancy, radiotherapy, or chemotherapy for malignancy (except BCC of the skin)
* Active autoimmune disease.
* Any past or present immunosuppressive treatment.
* Current treatment with chemotherapeutic agents
* History of metabolic bone disease (primary or secondary).
* Chronic renal insufficiency (defined by 50% increase of normal levels).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is to evaluate the proportion of infections at the treatment and control groups after six weeks | six weeks
  The primary endpoint of the study is to evaluate the proportion of infections at the treatment and control groups after six weeks

SECONDARY OUTCOMES:
1. To assess the proportion on infections at two weeks and 6 weeks of follow-up. | two weeks and six weeks
  To assess the proportion on infections at two weeks and 6 weeks of follow-up.
The number of patients recommended to undergo further procedural intervention because of the infection. | 12 MONTHS
  The number of patients recommended to undergo further procedural intervention because of the infection.